CLINICAL TRIAL: NCT03822546
Title: A Randomized, Open-label, Cross-over Clinical Study to Evaluate the Pharmacokinetic Profiles of Cigarettes and E-Cigarettes With Nicotine Salt Formulations in Adult Smokers
Brief Title: A Study to Evaluate the Pharmacokinetic Profiles of Cigarettes and E-Cigarettes With Nicotine Salt Formulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fontem Ventures BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: FON-01blu-2018
Record Dates: First submitted 2018-12-19; First posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Conventional cigarette (Experimental): The subject's preferred brand of commercially available conventional cigarette
  Interventions: Other: Conventional cigarette
- myblu 25 mg freebase (Active Comparator): myblu pod-system containing 25 mg nicotine ('freebase') tobacco flavour
  Interventions: Other: myblu 25 mg freebase
- myblu 16 mg nicotine salt (Active Comparator): myblu pod-system containing 16 mg nicotine salt tobacco flavour
  Interventions: Other: myblu 16 mg nicotine salt
- myblu 25 mg nicotine salt (Active Comparator): myblu pod-system containing 25 mg nicotine salt tobacco flavour
  Interventions: Other: myblu 25 mg nicotine salt
- myblu 40 mg nicotine salt (Active Comparator): myblu pod-system containing 40 mg nicotine salt tobacco flavour
  Interventions: Other: myblu 40 mg nicotine salt
- blu PRO 48 mg nicotine salt (Active Comparator): blu PRO open-system containing 48 mg nicotine salt tobacco flavour
  Interventions: Other: blu PRO 48 mg nicotine salt

INTERVENTIONS:
Other: Conventional cigarette — Subject's own conventional cigarette brand smoked with puffs taken at 30 seconds intervals
  Arms: Conventional cigarette
Other: myblu 25 mg freebase — E-cigarette used for 10 inhalations every 30 seconds
  Arms: myblu 25 mg freebase
Other: myblu 16 mg nicotine salt — E-cigarette used for 10 inhalations every 30 seconds
  Arms: myblu 16 mg nicotine salt
Other: myblu 25 mg nicotine salt — E-cigarette used for 10 inhalations every 30 seconds
  Arms: myblu 25 mg nicotine salt
Other: myblu 40 mg nicotine salt — E-cigarette used for 10 inhalations every 30 seconds
  Arms: myblu 40 mg nicotine salt
Other: blu PRO 48 mg nicotine salt — E-cigarette used for 10 inhalations every 30 seconds
  Arms: blu PRO 48 mg nicotine salt

SUMMARY:
This study evaluated the pharmacokinetic profiles and subjective effects of nicotine from two e-cigarette device platforms with varying concentrations of nicotine lactate (nicotine salt) e-liquid relative to conventional cigarettes. It was designed as a randomized, open-label, cross-over clinical study conducted in 15 healthy US adult smokers.

ELIGIBILITY:
Inclusion Criteria:

* Having smoked ≥10 manufactured cigarettes per day for at least the last year
* Expired carbon monoxide level of >10 ppm at screening
* Tested positive for urinary cotinine (≥500 ng/mL)

Exclusion Criteria:

* Known or suspected hypersensitivity to any component of the e-liquid formulations
* Taking or receiving prescription smoking cessation medicines
* Willing or considering to stop smoking
* Smokers who draw smoke into their mouth and throat but do not inhale
* Relevant illness history
* Body mass index (BMI) of less than 18 kg/m2 or greater than 40 kg/m2
* Breastfeeding women
* Women of child-bearing potential who were not using an accepted method of contraception

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Nicotine pharmacokinetics Cmax | 30 minutes following the start of product use (12 measurements over the period)
  Mean maximum plasma nicotine concentration (Cmax)
Nicotine pharmacokinetics Tmax | 30 minutes following the start of product use (12 measurements over the period)
  Median time to maximum plasma nicotine concentration (Tmax)
Nicotine pharmacokinetics AUC0-30 | 30 minutes following the start of product use (12 measurements over the period)
  Mean area under the plasma nicotine concertation-time curve, from time zero to 30 minutes (AUC0-30)

SECONDARY OUTCOMES:
Subjective effects questionnaire | 20 minutes after the start of product use
  Likert-type scale with responses ranging from 1 (not at all) to 7 (extremely). The following questions were asked: Did it make you dizzy? Did it make you nauseous? Did you enjoy it? Did it relieve the urge to smoke? Was it enough nicotine? Was it too much nicotine?
Incidence and nature of any adverse events (AE) | Through study completion, 6 days
  Incidence and nature of any adverse events (AE) (Safety and Tolerability)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No